CLINICAL TRIAL: NCT03278340
Title: Using Technology to Scale-Up an Occupational Sun Protection Policy Program
Acronym: SSW-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Kaiser Permanente (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0316; 0316 (Other: Klein Buendel, Inc.); R01CA210259 (NIH)
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Skin Cancer
Keywords: Skin Cancer; Prevention; Policy; Worksite; Scale-up; Cost and Effectiveness
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be aware of the condition in which their organization is assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sun Safe Workplaces - Technology (SSW-T) (Experimental): Program promoting the adoption of sun protection policies by fire departments and state Departments of Transportation that is delivered via a range of technology systems including web-enabled visits with senior managers, online training of outdoor workers, and online access to collateral materials (e.g., brochures, posters, tip cards).
  Interventions: Behavioral: Sun Safe Workplaces - Technology
- Sun Safe Workplaces - In Person (SSW-IP) (Active Comparator): Program promoting the adoption of sun protection policies by fire departments and state Departments of Transportation that is delivered via personal visits with senior managers and in person training of outdoor workers by research staff over two years. Collateral materials (e.g., brochures, posters, tip cards) will be provided to worksites.
  Interventions: Behavioral: Sun Safe Workplaces -In Person

INTERVENTIONS:
Behavioral: Sun Safe Workplaces - Technology — After randomization, program staff will contact managers at the recruited employer and schedule the initial web-enabled visit in the first 6 months. Follow-up meetings will be scheduled as needed to discuss policy adoption, and managers will schedule employee education using the SSW-T online training. Staff will follow-up with managers through Month 34 (Wave 1) or Month 46 (Wave 2). Electronic materials will be published on KB's state-of-the-art web server for employers to access and use.
  Other Names: SSW-T
  Arms: Sun Safe Workplaces - Technology (SSW-T)
Behavioral: Sun Safe Workplaces -In Person — After randomization, program staff will contact managers the recruited employer and schedule the initial in-person visit in the first 6 months. Follow-up meetings will be scheduled as needed to discuss policy adoption; managers will schedule employee education with SSW-IP project staff. Printed materials will be sent to SSW-IP employers 3 times during the intervention. Staff will follow-up with managers through Month 34 (Wave 1) or Month 46 (Wave 2).
  Other Names: SSW-IP
  Arms: Sun Safe Workplaces - In Person (SSW-IP)

SUMMARY:
Comprehensive approaches that combine sun protection policy and education for outdoor workers can reduce their risk for skin cancer by reducing their exposure to solar ultraviolet radiation on the job. To effectively disseminate the investigators' evidence-based sun protection policy and education intervention, Sun Safe Workplaces, a balance of effectiveness and cost of scale-up methods is required. The investigators propose to translate the intervention using a technology-based delivery method and compare the cost effectiveness of the original intervention and the intervention delivered by technology in a study that models national distribution strategies to public safety and public works sectors.

DETAILED DESCRIPTION:
A key goal in the Affordable Care Act is building a national culture of prevention through workplace health and safety initiatives. To achieve this goal, methods for scaling up evidence-based programs from research to wide-scale dissemination are needed to help balance effectiveness and cost. In many cases, there are pressures to reduce scale-up costs but at the expense of lower program implementation and effectiveness. A scale-up method that sacrifices effectiveness but reduces costs and reaches a larger number of employers may be acceptable. The investigators will model the effectiveness and cost trade-off, along with the extent and representativeness of reach, when scaling up the evidence-based occupational sun protection intervention, Sun Safe Workplaces (SSW), for national distribution. The intervention, which relies on personal contact with managers and in-person employee training (SSW-IP), created large improvements in comprehensive workplace sun safety (i.e., policy adoption and employee education) in a randomized controlled trial. The investigators will compare the existing in-person program delivery methods (SSW-IP) to a lower-cost dissemination method that utilizes Internet technology (SSW-T), i.e., virtual meetings, social networking, online training, and program materials. The aims of the research are to: 1) estimate the program reach (number and representativeness) and implementation rates (i.e., adoption of policies and delivery of education on occupational sun protection) achieved by the SSW-IP and SSW-T in a model of national distribution to public safety and public works industries; 2) estimate the costs associated with the SSW-IP and SSW-T (i.e., intervention costs and induced employer costs) and compare the estimated program benefits (i.e., policy and education) to cost; and 3) estimate the effect and cost-effectiveness of SSW-IP and SSW-T in secondary outcomes of a) changes in workplace environments and procedures for sun safety and b) workers' sun safety practices. In a 5-year project, SSW-T will be created by redesigning the very effective SSW-IP methods to use the latest web conferencing, social networking, and online training technology for dissemination. The implementation rates (defined as policy adoption and education delivery) and costs associated with SSW-IP (n=50 employers) and SSW-T (n=150 employers) will be modeled in a randomized two-group pretest-posttest design, enrolling a national sample of 200 employers (i.e., firefighting departments and state departments of transportation). Unlike traditional randomized trials, the primary analysis will be of cost effectiveness to test the hypothesis that SSW-T can be delivered cost-effectively to an expanded group of worksites producing a lower implementation rate than SSW-IP but at substantially lower cost. Secondary analyses will compare the two scale-up strategies on implementation rate, differences in rate by employer groups (e.g., size and region), changes to workplace environment/procedures, and employee sun safety practices. The findings will have high impact by helping public health practitioners select the best strategy for scaling up evidence-based workplace health and safety programs to achieve this ACA goal.

ELIGIBILITY:
Inclusion Criteria:

* Fire Departments and State DOTs in the United States, agreeing to participate, providing written policies at pretest and having at least 6 managers and 50 workers complete the pretest.
* Being a senior manager of a fire department or state DOT located in the United States. Criteria include a) being in a senior management position; b) responsible for work-site safety/health policy and education; c) consenting to participate, and d) completing the pretest. This includes city/county managers, human resources directors, risk managers, and managers of facilities, fire, roads and transportation departments
* Being an employee of a fire department or state DOT located in the United States. Criteria includes a) being employed part/full-time at the employer, b) working at least part of daytime hours outdoors, c) consenting to participate, and d) completing the pretest survey.

Exclusion Criteria:

* Prior participation in the Sun Safe Workplaces program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2644 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Implementation of Occupational Sun Protection Policy | Baseline to 2 years followup
  Policies will be collected from work sites and coded at both before and after the intervention period. Project staff will code written workplace policy documents on the presence of 15 "content categories" in three domains: 1) environmental controls; 2) administrative procedures; and 3) personal protection practices. Presence of policy is defined as having one or more policy components present in the written workplace policy documents (value = 1) versus no content components present (value = 0).
Implementation of Sun Safety Education | Baseline to 2 year followup
  Senior managers and employees will report on sun safety education provided to employees. The primary measure will be managers' reports of any training or any sun safety messages/materials distributed (e.g., newsletter articles, SSW website, or emails). Employees' reports of sun safety education will be secondary, validating managers' reports. These measures will be obtained in senior manager and employee pretest and posttest surveys, conducted online and by mail

SECONDARY OUTCOMES:
Economic Evaluation of the SSW-IP and SSW-T Intervention Programs | Baseline to 2 year followup
  Project staff will record costs associated with the SSW-IP and SSW-T, following protocols from prior projects. Project staff will identify resource allocations and both labor and non labor elements for each component of the SSW-IP and SSW-T (in-person and virtual visits; follow-up communications; staff-delivered and virtual training, web resources, and mailed materials). For personnel, the proportion of FTE across activities will be estimated by contemporaneous staff self-report. Senior manager and employee survey data will identify organizational changes induced by SSW-IP and SSW-T and attach cost estimates to each. The investigators will use the accounting systems of the trial itself, supplemented with survey responses and additional primary data collection or external sources. Costs will be recorded in custom-made spreadsheets and summed to produce overall cost estimates.
Changes in Workplace Environment for Sun Safety | Baseline to 2 year followup
  Managers will report changes in the work environments (providing shade and adjusting outdoor work schedules) or procedures (risk assessment, posting UV Index, and providing sunscreen, hats, protective clothing, and sunglasses) for sun safety. To validate, trained staff (blind to condition) will visit 18 randomly-selected employers at post-test and record shade, posting of UV Index, sunscreen availability, employee clothing, hats, and sunglasses, and educational materials, using a protocol from our Go Sun Smart trial.
Other Policy-related Measures | Baseline to 2 year followup
  The investigators will measure two ancillary policy outcomes in the senior manager surveys, the content of informal procedures (not written) and enforcement of any sun protection policies (i.e., how well is policy being implemented and how well are staff complying with policy [very well, well, about average, poorly, or very poorly]).
Employees Sun Protection Practices | Baseline to 2 year followup
  Employees will report a) frequency of sun protection at work, i.e., sunscreen with SPF 15+, long-sleeved shirts, long pants, hat with brim, sunglasses, shade use, limit exposure to midday sun, and have sunscreen, hat and eye protection at all times (1=never, 5=always) and b) prevalence of sunburn in the past three months on the job (yes/no; number of times) from SSW and GSS trials. These are standard, validated, and reliable measures from past studies.

CONTACTS AND LOCATIONS:
Overall Officials: David Buller, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - Kaiser Foundation Research Institute, Oakland, California
  - Klein Buendel, Inc., Golden, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buller DB, Buller MK, Meenan R, Cutter GR, Berteletti J, Eye R, Walkosz BJ, Pagoto S. Design and baseline data of a randomized trial comparing two methods for scaling-up an occupational sun protection intervention. Contemp Clin Trials. 2020 Oct;97:106147. doi: 10.1016/j.cct.2020.106147. Epub 2020 Sep 15. PMID 32942054